CLINICAL TRIAL: NCT04432649
Title: Multicenter Trial of Phase I/II Studies on CD276 (B7-H3) Positive Solid Tumors Treated With 4SCAR-276
Brief Title: Targeting CD276 (B7-H3) Positive Solid Tumors by 4SCAR-276
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Sun Yat-sen University (Other); Shenzhen Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20009
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effectiveness of 4SCAR-276 T cells (Experimental): The 4SCAR-276 T cells can recognize and kill tumor cells through the recognition of CD276 .This study will evaluate the side effects and effective doses of 4SCAR-276 T cells in treating refractory and recurrent solid tumors
  Interventions: Biological: 4SCAR-276

INTERVENTIONS:
Biological: 4SCAR-276 — The 4SCAR-276 T cells can recognize and kill tumor cells through the recognition of CD276 .This study will evaluate the side effects and effective doses of 4SCAR-276 T cells in treating refractory and recurrent solid tumors
  Other Names: CD276-specific 4th Generation CART

SUMMARY:
Patients with refractory and/or recurrent solid tumor have poor prognosis despite complex multimodel therapy and therefore, novel approaches are urgently needed. This study attempts to treat these diseases using T cells genetically modified with a 4th generation lentiviral chimeric antigen receptor (4SCAR fused with an inducible apoptotic caspase 9 domain) targeting CD276 (B7-H3). The 4SCAR-CD276-modified T cells (4SCAR-276) can recognize and kill tumor cells through the recognition of CD276, a surface protein expressed at high levels on many types of tumors but at low levels on normal tissues. This study will evaluate the side effects and effective doses of 4SCAR-276 in treating refractory and/or recurrent tumors.

DETAILED DESCRIPTION:
Background: Patients with refractory and/or recurrent solid tumors have poor prognosis despite complex multimodal therapy; therefore, novel curative approaches are needed. The investigators are attempting to use T cells obtained directly from the patient, which can be genetically modified to express a 4th generation CD276-specific chimeric antigen receptor (4SCAR-276). The CAR molecules enable the T cells to recognize and kill tumor cells through the recognition of the surface CD276, which is expressed at high levels on tumor cells including brain tumors, Ewing's sarcoma (PNET) and many other tumors but not at significant levels on normal tissues. This study will evaluate the side effects and the best dose of a novel 4th generation anti-CD276 CAR T cells to target refractory and/or recurrent solid tumors.

Design:

1. Participants will be screened through physical exam and medical history. Blood and tumor tissue samples will be collected. Imaging studies will be performed.
2. Peripheral blood mononuclear cells (PBMC) will be obtained by apheresis, and T cells will be activated and modified to express the 4SCAR-276 gene.
3. On Day -5 to -7, PBMC will be activated and enriched for T cells, which will be followed by 4SCAR-276 lentiviral transduction. The total culture time is approximately 5-7 days.
4. Participants will receive a preparative conditioning regimen comprising cyclophosphamide/fludarabine to prepare their immune system to accept the modified CAR T cells. The preparative regimen will be based on patient immune condition and consistent with standard chemotherapy conditioning regimen.
5. The patients will receive ~10^6 CART cells/kg body weight per infusion, and may receive additional booster CART infusions if positive outcome is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors have received standard first-line therapy and have been judged to be non-resectable, metastatic, progressive or recurrent.
* The CD276 antigen status of the tumor is determined for eligibility. Positive expression is defined by antibody staining results based on immunohistochemistry or flow cytometry analysis.
* Body weight greater than or equal to 10 kg.
* Age: ≥1 year and ≤ 75 years of age at the time of enrollment.
* Life expectancy: at least 8 weeks.
* Prior Therapy: 1) There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less. 2) Must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection. 3) At least 7 days must have elapsed since the completion of therapy with a biologic agent, targeted agent, tyrosine kinase inhibitor or a metronomic nonmyelosuppressive regimen. 4) At least 4 weeks must have elapsed since prior therapy that included a monoclonal antibody. 5) At least 1 week since any radiation therapy at the time of study entry.
* Karnofsky/jansky score of 60% or greater.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent .
* Pulse Ox greater than or equal to 90% on room air.
* Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
* Renal function: Patients must have serum creatinine less than 3 times upper limit of normal.
* Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease not evaluable to have hematologic toxicity.
* For all patients enrolled in this study, themselves or their parents or legal guardians must sign an informed consent and assent.

Exclusion Criteria:

Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, or grade 3 hematologic toxicity.

* Untreated central nervous system (CNS) metastasis: Patients with CNS tumor involvement that has been treated and/or is stable for at least 6 weeks following completion of therapy are eligible.
* Previous treatment with other genetically engineered CD276-CAR T cells or CD276 antibody therapy.
* Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
* Patients who require systemic corticosteroid or other immunosuppressive therapy.
* Evidence of tumor potentially causing airway obstruction.
* Inability to comply with protocol requirements.
* Insufficient CAR T cells availability.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 3 years
  Determine the toxicity profile the 4SCAR-276-modified T cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 1 year
  Defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) based on imaging analysis.
Survival time of the patients | 3 years
  Evaluate the survival time of the patients treated with the 4SCAR-276 T cells, including progression free survival (PFS) and overall survival (OS).

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Sun Yat-Sen University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No